CLINICAL TRIAL: NCT05344937
Title: Estudio de validación de Uromonitor en el diagnóstico Precoz de cáncer Vesical en Pacientes de Alto Riesgo Con Microhematuria
Brief Title: Validation Study of Uromonitor in High Risk Microhematuria Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Collaborators: IPATIMUP - Instituto De Patologia E Imunologia Molecular Da Universidade Do Porto (Other)
Responsible Party: Sponsor
Other Study IDs: UROSCAVCUN
Record Dates: First submitted 2022-04-19; First posted 2022-04-25 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Biospecimen Retention: Samples With DNA — Urine DNA
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Men over 40 years of age, and women over 50, smokers or former smokers with a smoking rate greater than 10 packs/year and the presence of microhematuria >25 red blood cells per field in the microscopic analysis are at high risk of bladder cancer, so cystoscopy and uroTAC is advised in the AUA Guidelines.

The investigators hypothesize if cystoscopy can be omitted in case of having a negative biomarker test and a normal uro-CT.

Main objective: To determine sensitivity, specificity, positive and negative predictive value of "Uromonitor" (molecular DNA based urine marker) in the included population, in relation to the presence of urothelial cancer in the bladder, comparing it with cystoscopy.

DETAILED DESCRIPTION:
1. Title: Validation study of Uromonitor in the early diagnosis of bladder cancer in high-risk patients with microhematuria. Version: 2.0. March 6, 2022.

   Main author: Felipe Villacampa Aubá. Department of Urology, University Clinic of Navarra (CUN).
2. Justification and context. Patients with microhematuria and smokers have a high risk of having bladder cancer (5-10%), so a cystoscopy and Urotac should be performed.

   Cystoscopy is an uncomfortable test, which is rejected by many patients. The aim is to assess whether a urine molecular marker, already validated in other situations, is capable of substituting cystoscopy, improving the study of these patients and avoiding uncomfortable and invasive diagnostic tests for the patient.
3. Hypotheses and research objectives. Hypothesis: Men over 40 years of age, and women over 50, smokers or ex-smokers with a smoking rate greater than 10 packs/year and the presence of microhematuria >25 red blood cells per field in the microscopic analysis (high risk) can omit cystoscopy in case of having a negative biomarker test and a normal uro-CT.

   Main objective: To determine sensitivity, specificity, positive and negative predictive value of "Uromonitor" in the included population, in relation to the presence of urothelial cancer in the bladder, comparing it with cystoscopy.
4. Study design. This is a prospective observational study, in which the results of the "Uromonitor" test in urine are compared with the results of cystoscopy, a standard test in the population studied, to be able to detect urothelial cancer in the bladder.

   Patients seen at the University Clinic of Navarra by the Neurology Department (Pamplona and Madrid) with microhaematuria of more than 25 red blood cells per field will be included, being referred to urology department to study the risk of bladder cancer.

   There is the possibility of expanding the study to a center in Portugal with the same inclusion and exclusion criteria and the same protocol. This management is being carried out and will be confirmed throughout the study.
5. Population. Population studied for opportunistic screening in lung cancer, which, if presenting a urine sediment with more than 25 red cells hps, is considered to be at high risk for bladder cancer according to the guidelines of the American Urological Association (AUA) of 2020.
6. Variables.

   * Age
   * Sex
   * Date of birth
   * Smoking status (active smoker, ex-smoker)
   * Smoking rate
   * Red blood cells by field in microscopic analysis of urine
   * CT results
   * Urine cytology results
   * Cystoscopy results
   * Uromonitor results
   * Date of bladder TUR (if carried out)
   * Date of nephroureterectomy (if carried out)
   * Result of pathological anatomy (in case of biopsy or surgery)
   * Final diagnosis.
7. Data sources. For the clinical variables, the usual medical records will be used. For the results of the uromonitor, the results sent by the manufacturer will be used.
8. Study size. Assuming a prevalence of 7%, an expected sensitivity and specificity of 90%, and considering a confidence of 95% and a clinically acceptable precision of 12%, a sample size required for the study of 343 patients is estimated.
9. Data analysis. Quantitative clinical and demographic variables will be described by mean and standard deviation. Qualitative variables will be described by absolute and relative distribution frequencies. The sensitivity, specificity, positive predictive value and negative predictive value of the test under evaluation will be estimated, with their respective 95% confidence intervals. Statistical analyzes will be performed using Stata software (StataCorp. 2015. Stata Statistical Software: Release 14. College Station, TX: StataCorp LP).

ELIGIBILITY:
Inclusion Criteria (all conditions must be certified):

* Men over 40 years of age or Women over 50 years of age.
* Smokers or former smokers
* Smoking rate >10 packs/year
* Microhematuria with >25 red blood cells per hpf.

Exclusion Criteria: (any of them):

* Patients who refuse to undergo cystoscopy.
* Patients who refuse or cannot perform imaging tests of the upper section due to allergy or chronic kidney disease.
* History of macroscopic hematuria.
* History of microscopic hematuria already known and studied.
* Known cause of microhematuria: e.g. urinary infection, bladder lithiasis
* Patients who refuse to participate in the study.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Men and women seen for being at risk of lung cancer are included, and who present microhematuria above 25 red blood cells per field, so they are also at high risk for bladder cancer.
Sampling Method: Non-Probability Sample
Enrollment: 343 (Estimated)
Dates: Start 2022-05-02 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Accuracy of Uromonitor in diagnosis of bladder cancer in high risk micro hematuria | 18 months
  Specificity, sensibility, negative and positive predictive value of Uromonitor in high risk microhematuria patients

SECONDARY OUTCOMES:
acuracy of Uromonitor in diagnosis of high grade bladder tumours in this population | 18 months
  Sensibility of uromonitor in detecting high grade bladder tumours

CONTACTS AND LOCATIONS:
Overall Officials: Felipe Villacampa, MD, Principal Investigator — Clinica Universidad de Navarra
Locations (1):
- Clinica Universidad de Navarra, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Barocas DA, Boorjian SA, Alvarez RD, Downs TM, Gross CP, Hamilton BD, Kobashi KC, Lipman RR, Lotan Y, Ng CK, Nielsen ME, Peterson AC, Raman JD, Smith-Bindman R, Souter LH. Microhematuria: AUA/SUFU Guideline. J Urol. 2020 Oct;204(4):778-786. doi: 10.1097/JU.0000000000001297. Epub 2020 Jul 23. PMID 32698717
- [Background] Laukhtina E, Shim SR, Mori K, D'Andrea D, Soria F, Rajwa P, Mostafaei H, Comperat E, Cimadamore A, Moschini M, Teoh JY, Enikeev D, Xylinas E, Lotan Y, Palou J, Gontero P, Babjuk M, Witjes JA, Kamat AM, Roupret M, Shariat SF, Pradere B; European Association of Urology-Young Academic Urologists (EAU-YAU): Urothelial Carcinoma Working Group. Diagnostic Accuracy of Novel Urinary Biomarker Tests in Non-muscle-invasive Bladder Cancer: A Systematic Review and Network Meta-analysis. Eur Urol Oncol. 2021 Dec;4(6):927-942. doi: 10.1016/j.euo.2021.10.003. Epub 2021 Nov 6. PMID 34753702
- [Background] Sieverink CA, Batista RPM, Prazeres HJM, Vinagre J, Sampaio C, Leao RR, Maximo V, Witjes JA, Soares P. Clinical Validation of a Urine Test (Uromonitor-V2(R)) for the Surveillance of Non-Muscle-Invasive Bladder Cancer Patients. Diagnostics (Basel). 2020 Sep 24;10(10):745. doi: 10.3390/diagnostics10100745. PMID 32987933